CLINICAL TRIAL: NCT06875895
Title: Effect of Motor Imagery Training on Pain, Functionality, Proprioception and Kinesiophobia in Patients With Partial Rotator Cuff Tears
Brief Title: Effect of Motor Imagery Training on Pain, Functionality, Proprioception and Kinesiophobia in Partial Rotator Cuff Tear
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevtap Cakir, Asst. Prof., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSBU-RC
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator Cuff; Exercise therapy; Imagery
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: A single-center randomized controlled study was designed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Traditional Physiotherapy) (Active Comparator): Traditional physical therapy will begin with the application of Hotpack, Tens and Ultrasound to the painful area for five minutes. Then, stretching exercises will be performed at the pain limit for the six main shoulder movements in the shoulder joint. Then, wand exercises, pendulum exercises, isometric exercises for the shoulder joint and strengthening active exercises will be given in order to increase the normal range of motion in the shoulder joint. The six main shoulder movements will be actively performed (flexion, extension, abduction, adduction, medial and lateral rotations). After the 5th session, weights will be added according to the patient's condition.
  Interventions: Other: Traditional Physiotherapy
- Motor Imagery Training (Experimental): In motor imagery training, exercises in traditional physiotherapy will be applied with kinesthetic and visual motor imagery. Each movement will be divided into five sets consisting of two trials separated by 10 repetitions and 30-second rest periods. It will also be emphasized through practice that the functional movement imagined and the times when this movement is actually actively performed should be similar. Individuals' eyes will be closed throughout the entire motor imagery training. At the very beginning of the session, a relaxation exercise lasting approximately 5 minutes will be performed in order to maximize attention during motor imagery. Whether or not individuals are performing imagery will be monitored by monitoring heart rate variables from autonomic functions. In order to ensure standardization during imagery, commands will be applied with audio recordings containing metaphors.
  Interventions: Other: Motor Imagery Training

INTERVENTIONS:
Other: Traditional Physiotherapy — Hotpack, Tens and Ultrasound application
  Arms: Control Group (Traditional Physiotherapy)
Other: Motor Imagery Training — Kinesthetic and visual motor imagery will be applied.
  Arms: Motor Imagery Training

SUMMARY:
The aim of this study is to investigate the effects of motor imagery training on pain, functionality, proprioception and kinesiophobia in patients with partial rotator cuff tears. Participants will be randomly assigned to traditional physiotherapy and motor imagery groups. Interventions will be performed with a physiotherapist for a total of 20 sessions for 4 weeks, 5 days a week. The intervention program will be determined by the Specialist Physical Therapy Physician. Data will be collected before the study, at the end of the training in the 4th week and at the 8th week (follow-up evaluation). Motor imagery ability will be assessed with the Movement Imagery Questionnaire (MIQ-R), pain will be assessed with the Numerical Assessment Scale for functionality with the DASH, proprioception will be assessed with the inclinometer and kinesiophobia will be assessed with the Tampa Kinesiophobia Scale.

DETAILED DESCRIPTION:
One of the most common pathologies related to the shoulder joint, which has a wide range of motion, is the tears of varying degrees in the rotator cuff muscles. The rotator cuff muscles consist of the dynamic stabilizers of the shoulder: supraspinatus, infraspinatus, subscapularis and teres minor muscles. Pathologies related to the rotator cuff can present as simple overuse, impingement syndrome, partial tear, full-thickness tear and, in the advanced stage of the tear, rotator cuff tear arthropathy. Such tears can usually occur due to injuries and traumas, degeneration due to aging, overuse or repetitive movements. The main symptoms of a partial rotator cuff tear are increased shoulder pain during overhead movements, limited movement, muscle weakness and loss of function. Partial rotator cuff tear is usually diagnosed with physical examination and imaging techniques such as MRI (Magnetic Resonance Imaging), ultrasonography, and X-ray. The treatment approach varies depending on the size of the tear, the patient's symptoms, and lifestyle, and is divided into conservative treatments and surgical techniques. Motor imagery is the individual's conscious simulation of the movement without any motor output. Motor imagery contributes to the improvement of motor performance and the learning of new motor skills. Motor imagery is divided into two as visual and kinesthetic imagery. While visual imagery consists of visualizing the movement, kinesthetic imagery focuses on the position of the muscles and limbs and the somatic sensations created by their movement. Studies combining motor imagery with classical physiotherapy training show that it increases the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Partial rotator cuff tear diagnosis.
* Between the ages of 18-65
* Patients experiencing pain for at least 4 weeks.
* Having a valid score on the Mini Mental Test (>24)
* Those without a history of any neurological or serious psychological illness.
* Those who have not participated in a previous study on motor imagery training

Exclusion Criteria:

* Complete rotator cuff tear or conditions requiring surgical intervention,
* Participants who have received treatment with corticosteroids by any means in the previous 6 months,
* Participants who have a rotator cuff tear due to acute traumatic conditions (proximal humerus fracture).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Randomization was done according to gender, 40 female and 40 male.
Enrollment: 80 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Standardized Mini Mental Test | a day before the rehabilitation
  The Standardized Mini Mental Test is a short, efficient and standard method that can be preferred in determining the cognitive level of the individual. It is collected under five headings: orientation, recording memory, attention and calculation, recall and language. There are eleven items that individuals will answer. It is evaluated out of a total of 30 points. The threshold value was determined as 24 points in the Turkish validity and reliability study.
Numerical Rating Scale | a day before the rehabilitation
  Pain intensity will be measured using the Numerical Rating Scale. A decrease in the point indicates that the pain is decreasing.
Numerical Rating Scale | up to 4 weeks
  Pain intensity will be measured using the Numerical Rating Scale. A decrease in the point indicates that the pain is decreasing.
Numerical Rating Scale | up to 8 weeks
  Pain intensity will be measured using the Numerical Rating Scale. A decrease in the point indicates that the pain is decreasing.
Disabilities of the arm, shoulder, and hand | a day before the rehabilitation
  Disabilities of the arm, shoulder, and hand scale is a questionnaire developed to assess the musculoskeletal pathology of the upper extremity and the entire upper extremity in general. It consists of 30 questions that evaluate the degree of difficulty in performing different activities using the upper extremity in daily life in the last week (21 questions), symptoms consisting of pain, activity-related pain, numbness, joint stiffness and weakness (5 questions), and the effects of pathologies on social life, sleep, work and psychological status (4 questions). All questions have a 5-point Likert model (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: completely unable to do). The Turkish version of the DASH Questionnaire was used.
Disabilities of the arm, shoulder, and hand | up to 4 weeks
  Disabilities of the arm, shoulder, and hand scale is a questionnaire developed to assess the musculoskeletal pathology of the upper extremity and the entire upper extremity in general. It consists of 30 questions that evaluate the degree of difficulty in performing different activities using the upper extremity in daily life in the last week (21 questions), symptoms consisting of pain, activity-related pain, numbness, joint stiffness and weakness (5 questions), and the effects of pathologies on social life, sleep, work and psychological status (4 questions). All questions have a 5-point Likert model (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: completely unable to do). The Turkish version of the DASH Questionnaire was used.
Disabilities of the arm, shoulder, and hand | up to 8 weeks
  Disabilities of the arm, shoulder, and hand scale is a questionnaire developed to assess the musculoskeletal pathology of the upper extremity and the entire upper extremity in general. It consists of 30 questions that evaluate the degree of difficulty in performing different activities using the upper extremity in daily life in the last week (21 questions), symptoms consisting of pain, activity-related pain, numbness, joint stiffness and weakness (5 questions), and the effects of pathologies on social life, sleep, work and psychological status (4 questions). All questions have a 5-point Likert model (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: completely unable to do). The Turkish version of the DASH Questionnaire was used.
Tampa Kinesiophobia Scale | a day before the rehabilitation
  The Tampa Kinesiophobia Scale will be used. A 4-point Likert scale is used and the total score is 33. The higher a person's score on the scale, the greater their fear of movement.
Tampa Kinesiophobia Scale | up to 4 weeks
  The Tampa Kinesiophobia Scale will be used. A 4-point Likert scale is used and the total score is 33. The higher a person's score on the scale, the greater their fear of movement.
Tampa Kinesiophobia Scale | up to 8 weeks
  The Tampa Kinesiophobia Scale will be used. A 4-point Likert scale is used and the total score is 33. The higher a person's score on the scale, the greater their fear of movement.

SECONDARY OUTCOMES:
Movement Imagery Questionnaire (MIQ-R) | a day before the rehabilitation
  This is an 8-item self-report questionnaire in which participants rate the vividness of their mental representations using a 7-point scale (1 = very difficult to see/feel and 7 = very easy to see/feel). This test will be used to ensure that the sample does not include individuals with extremely high or low motor imagery ability
Movement Imagery Questionnaire (MIQ-R) | up to 4 weeks
  This is an 8-item self-report questionnaire in which participants rate the vividness of their mental representations using a 7-point scale (1 = very difficult to see/feel and 7 = very easy to see/feel). This test will be used to ensure that the sample does not include individuals with extremely high or low motor imagery ability
Movement Imagery Questionnaire (MIQ-R) | up to 8 weeks
  This is an 8-item self-report questionnaire in which participants rate the vividness of their mental representations using a 7-point scale (1 = very difficult to see/feel and 7 = very easy to see/feel). This test will be used to ensure that the sample does not include individuals with extremely high or low motor imagery ability

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)